CLINICAL TRIAL: NCT04426240
Title: A Comparative Study of Use of Cyclosporin Eye Before Cataract Surgery for the Prevention of Dry Eye
Brief Title: The Effect of Cyclosporin Before Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, tae-young chung, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-11-203
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclosporine (Active Comparator): Subject who use cyclosporine and hyaluronate artificial tear 1 month before cataract surgery
  Interventions: Drug: Cyclosporine microemulsion
- non-Cyclosporine (No Intervention): Subject who use only hyaluronate eye drop 1 month before cataract surgery

INTERVENTIONS:
Drug: Cyclosporine microemulsion — Intervention group receives topical cyclosporine dry eye treatment before cataract surgery
  Other Names: Cyporin
  Arms: Cyclosporine

SUMMARY:
To evaluate the effect of cyclosporine eye drop before cataract surgery for the prevention of post cataract surgery dry eye syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. 21+ adult men and women
2. Those who are scheduled to undergo cataract surgery due to a diagnosis of cataract
3. Corneal fluorescein staining score (Oxford) is II or less
4. Preoperative MMP-9 positive
5. Those who have not used the trial and the test (cyclosporine) for at least 1 month before surgery.
6. Those who have voluntarily written consent to participate in this clinical trial

Exclusion Criteria

1. Those who have used systemic or topical cyclosporine within 4 weeks
2. Use of eye drops for more than 4 weeks (disorders, allergies, eye inflammation / infection, etc.) other than the current dry eye syndromes
3. Patients who have systemic or ocular disorders or conditions (eye surgery, trauma, disease) that can influence the results of this trial.
4. Abnormal eyelid function
5. An eye disease that can impair the function of the corneal sensation: herpes keratopathy, conjunctival wounds due to scarring conjunctivitis, pterygium, pinguecula, diabetic keratitis, keratoconus , corneal transplant status
6. Patients with active eye infections
7. Patients with conflicts with this clinical trial
8. Pregnant and lactating mothers
9. Patients who are determined to be inappropriate by other investigators

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Corneal florescence staining score | 1 month
  Standardized corneal staining score (NEI score, National eye institute score) : dividing the cornea into five sections and assigning a value from 0 (absent) to 3 (severe) to each section, based on the amount, size, and confluence of the PEE, for a maximum of 15 points.

SECONDARY OUTCOMES:
tear break-up time | 1 month
  Time to break tear film
Schirmer test | 1 montn
  Tear secretion test

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Young Chung, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea